CLINICAL TRIAL: NCT00924807
Title: Phase I/II Study of Sorafenib Concurrent With Androgen Deprivation and Radiotherapy in the Treatment of Intermediate- and High-Risk Localized Prostate Cancer
Brief Title: Safety Study of Sorafenib With Androgen Deprivation and Radiotherapy to Treat Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor closed the trial
Sponsor: Beth Israel Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 004-08; SR06-959
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Combined Androgen Blockade; Radiotherapy; Sorafenib
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; bicalutamide; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Androgen Depr, Radiotherapy, Sorafenib (Experimental): Everyone will receive Leuprolide acetate, Bicalutamide,Sorafenib and radiotherapy.
  Interventions: Drug: Leuprolide acetate, Bicalutamide, Sorafenib

INTERVENTIONS:
Drug: Leuprolide acetate, Bicalutamide, Sorafenib — Leuprolide acetate - depot, Bicalutamide 50 mg, Sorafenib 400mg
  Other Names: Leuprolide acetate; Bicalutamide; Sorafenib

SUMMARY:
The purpose of this study is to evaluate the safety of a new drug- sorafenib, which is to be administered at the same time as standard treatment, which includes hormonal therapy and external beam radiotherapy.

DETAILED DESCRIPTION:
Leuprolide acetate (a luteinizing hormone releasing hormone (LHRH) agonist) and Bicalutamide (an anti-androgen) are hormonal agents which are commonly used to reduce testosterone blood level for prostate cancer treatment. Intensity modulated external beam radiotherapy is a standard treatment for localized prostate cancer. Previous studies have shown that combining hormonal therapy and radiation is more effective than radiation alone. Unfortunately, significant percentages (50-75%) of patients still relapse. Sorafenib reduces the growth of cancer cells and has proven effective in the treatment of solid tumors including kidney and liver cancer. This drug is approved by the FDA for treatment kidney and liver cancer. The study investigators believe that adding sorafenib to standard treatment, comprising hormonal therapy and radiation, might be more effective then standard hormonal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed intermediate or high risk prostate adenocarcinoma. Intermediate risk disease comprises T2b/c tumors, Gleason 7 histology, or PSA 10-20. High risk tumors comprise T3-4, Gleason 8 or higher histology, or PSA greater than 20.
* Age > 18 years.
* Life expectancy of greater than 5 years.
* Patients must have normal organ and marrow function.
* No pelvic lymph node metastases based on pelvic CT scan or MRI.
* No bone metastasis. A whole body bone scan is required to rule out metastatic disease.

Exclusion Criteria:

* Any previous, radiotherapy, or chemotherapy, or more than 4 weeks of androgen deprivation hormonal therapy for the treatment of prostate adenocarcinoma.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib or other agents used in this study.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin will not be allowed to participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Cohen, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St.Luke's-Roosevelt Hospital Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Androgen Depr, Radiotherapy, Sorafenib
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Androgen Depr, Radiotherapy, Sorafenib
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 66.25 [61 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 4
Gleason 7 histology, or PSA 10-20 [Number; unit: participants] — Prostate cancers are commonly graded using Gleason score or pattern. Gleason grading is based on a 5-component system, based on 5 histologic patterns.
  Cancers with a Gleason score of 7 may be called moderately differentiated or intermediate grade.
  Prostate-Specific Antigen (PSA) a protein that is produced by the prostate gland. The higher a man's PSA level, the more likely it is that he has prostate cancer. Most doctors considered PSA levels of 4.0 ng/mL and lower as normal.
  participants | 4

OUTCOME MEASURES:

1. Primary Outcome: Determine the Safety and Maximally Tolerated Dose of Sorafenib Administered Concurrently With Radiotherapy in the Treatment of Intermediate- and High-risk Localized Prostate Cancer.
Description: Data of zero ("0") participants were analyzed due to lack of funding and prematurely terminating the study by sponsor. All subjects are following up in the clinic off the study.
Time Frame: Day 29 and every 2 weeks
Population: Data of zero ("0") participants were analyzed due to lack of funding and prematurely terminating the study by sponsor. All subjects are following up in the clinic off the study.
Arm/Group | Androgen Depr, Radiotherapy, Sorafenib
Number analyzed (Participants) | 0

2. Secondary Outcome: Biochemical Disease-free Survival
Description: as for outcome 1
Time Frame: after 9 months
Population: data not collected
Arm/Group | Androgen Depr, Radiotherapy, Sorafenib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 18 months
Description: Adverse Events were assessed by regular investigator assessment, regular laboratory testing
Arm/Group | Androgen Depr, Radiotherapy, Sorafenib
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Androgen Depr, Radiotherapy, Sorafenib (N=4)
Hypertension (Cardiac disorders) | 3 (3)
Urinary frequency/urgency (Renal and urinary disorders) | 4 (4)
Urinary retention (Renal and urinary disorders) | 1 (1)
dysuria (Renal and urinary disorders) | 3 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Hot flashes (Endocrine disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2)
Proctitis (Gastrointestinal disorders) | 1 (1)
Ocular-Amaurosis fugax (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Data of zero ("0") participants were analyzed due to lack of funding and prematurely terminating the study by sponsor. All subjects are following up in the clinic off the study. Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes